CLINICAL TRIAL: NCT01132625
Title: A Japanese Phase I, Multi-center, Open-label, Study of AUY922 Administered Intravenously on a Once Weekly Schedule in Adult Patients With Advanced Solid Malignancies
Brief Title: Dose Escalation Study of AUY922 in Advanced Solid Malignancies in Japan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAUY922A1101
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2013-02

CONDITIONS: Advanced Solid Tumors
Keywords: HSP90; molecular chaperone; advanced solid tumors; Japan
MeSH Terms: interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide

ARMS (1):
- AUY922 (Experimental)
  Interventions: Drug: AUY922

INTERVENTIONS:
Drug: AUY922

SUMMARY:
This study will characterize the safety, tolerability, efficacy, pharmacokinetics, and pharmacodynamics of AUY922 in adult patients with advanced solid malignancies in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced malignant solid tumors
* ECOG Performance Status of ≤ 2
* Patients must have the following laboratory values:
* Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L, Hemoglobin (Hgb) ≥ 8.5 g/dl, Platelets (plt) ≥ 100 x 109/L
* Potassium, Calcium, Magnesium, Phosphorus within normal limits or correctable with supplements
* AST/SGOT and ALT/SGPT ≤ 2.5 x Upper Limit of Normal (ULN)
* Serum bilirubin ≤ 1.5 x ULN, Serum albumin > 2.5g/dl, Serum creatinine≤ 1.5 x ULN or 24-hour clearance ≥ 50 ml/min
* Able to sign informed consent and to comply with the protocol

Exclusion Criteria:

* Patients with brain metastasis.
* Prior treatment with any HSP90 or HDAC inhibitor compound.
* Treatment with therapeutic doses of coumarin anticoagulants.
* Pregnant and lactating women.
* Severe and/or uncontrolled acute or chronic liver disease
* Severe and/or uncontrolled acute or chronic renal disease
* Chronically significant heart disease
* History (or family history) of long QT syndrome. QTc ≥ 450 msec on screening ECG, ischemic heart disease, heart fail, ECG abnormalities, atrial fibrillation, atrial flutter or ventricular arrhythmias including ventricular tachycardia or Torsades de Pointes.
* Patients who are currently receiving treatment with any medication which has a relative risk or prolonging the QTcF interval or inducing Torsades de Pointes
* Patients with known disorders due to a deficiency in bilirubin glucuronidation (e.g Gilbert's syndrome).

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
establish maximum tolerate dose (safety and tolerability) | about 3 years

SECONDARY OUTCOMES:
Safety assessed by type, frequency and severity of adverse events | about 4 years
Efficacy assessed by RECIST | about 4 years
Pharmacokinetic assessed by Cmax, Tmax, AUC | about 3 years
Pharmacodynamic assessed by blood and tumor biomarkers at baseline and post AUY922 | about 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Japan (2):
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Sunto-gun, Shizuoka

REFERENCES:
- See also: Results for CAUY922A1101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=8084